CLINICAL TRIAL: NCT00759395
Title: An Investigation of the Antidepressant Efficacy of a Selective, High, Affinity Enkephalinergic Agonist in Anxious Major Depressive Disorder
Brief Title: Study of Antidepressant Efficacy of a Selective, High Affinity Enkephalinergic Agonist in Anxious Major Depressive Disorder (AMDD)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: D0880C00021; NCT00738270 (obsolete NCT alias)
Record Dates: First submitted 2008-09-24; First posted 2008-09-25 (Estimated); Results first posted 2012-11-08 (Estimated); Last update posted 2012-11-08 (Estimated); Status verified 2012-10

CONDITIONS: Anxious Major Depressive Disorder
Keywords: Anxious Major Depressive Disorder
MeSH Terms: interventions — 4-((3-aminophenyl)(4-(4-fluorobenzyl)piperazin-1-yl)methyl)-N,N-diethylbenzamide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- AZD2327 (Experimental): AZD2327 3mg BID
  Interventions: Drug: AZD2327
- Placebo (Placebo Comparator): Placebo BID
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AZD2327 — Tablet, Oral, Daily
  Arms: AZD2327
Drug: Placebo — Tablet, Oral, Daily
  Arms: Placebo

SUMMARY:
This study will determine if a highly selective enkephalinergic receptor modulator is effective in the treatment of anxious major depressive disorder.

ELIGIBILITY:
Inclusion Criteria:

* Provision of informed consent prior to any study specific procedures
* Diagnosis of major depressive disorder without psychotic features (MDD)

Exclusion Criteria:

* A history of substance or alcohol abuse within the past 6 months or dependence within 1 year of enrollment as defined by DSM-IV criteria.
* Women that are pregnant or lactating
* History of pancreatitis

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2009-01; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Smith, MD, Study Director — AstraZeneca; Carlos Zarate, Principal Investigator — National Institute of Mental Health (NIMH)
Locations (1):
- Research Site, Baltimore, Maryland, United States

REFERENCES:
- [Derived] Richards EM, Mathews DC, Luckenbaugh DA, Ionescu DF, Machado-Vieira R, Niciu MJ, Duncan WC, Nolan NM, Franco-Chaves JA, Hudzik T, Maciag C, Li S, Cross A, Smith MA, Zarate CA Jr. A randomized, placebo-controlled pilot trial of the delta opioid receptor agonist AZD2327 in anxious depression. Psychopharmacology (Berl). 2016 Mar;233(6):1119-30. doi: 10.1007/s00213-015-4195-4. Epub 2016 Jan 4. PMID 26728893

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A single site, randomized, double blind, placebo-controlled, parallel group experimental study. Patients recruited between November 2008 and October 2011.
Pre-assignment Details: Screening for eligibility and wash-out of restricted medications.
Groups:
- AZD2327: AZD2327 3mg BID Tablet, Oral, Daily
- Placebo: Placebo BID, Tablet, Oral, Daily
Period: Overall Study
Arm/Group | AZD2327 | Placebo
Started | 13 | 9
Completed | 11 | 7
Not Completed | 2 | 2
Not completed — Adverse Event | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Lack of Efficacy | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | AZD2327 | Placebo | Total
Number analyzed (Participants) | 13 | 9 | 22
Age Continuous [Mean (Standard Deviation); unit: Years] | 40 (12.2) | 48.7 (11.3) | 44.35 (11.75)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 5 | 12
  Male | 6 | 4 | 10

OUTCOME MEASURES:

1. Primary Outcome: Hamilton Rating Scale for Depression (HAM-D) Total Score.
Description: Hamilton Rating Scale for Depression (HAM-D)is a 17-item, clinician-rated scale that assesses depressive symptoms. The HAMD-17 consists of 17 symptoms, each of which is rated from 0 to 2 or 0 to 4, where 0 is none/absent. The HAMD-17 total score is calculated as the sum of the 17 individual symptom scores; the total score can range from 0 to 52. Higher HAMD-17 scores indicate more severe depression.
Time Frame: Week 4
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | AZD2327 | Placebo
Number analyzed (Participants) | 13 | 9
Units on a scale | 14.249 (2.152) | 16.307 (2.604)

2. Primary Outcome: Hamilton Rating Scale for Anxiety (HAM-A) Total Score.
Description: The Hamilton Rating Scale for Anxiety (HAM-A) is used as a rating measure of anxiety severity. The scale consists of 14 items. Each item is rated on a scale of 0 to 4. The HAM-A total score is the sum of the 14 items and the score ranges from 0 to 56, 0 is considered the best outcome.
Time Frame: Week 4
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | AZD2327 | Placebo
Number analyzed (Participants) | 13 | 9
Units on a scale | 13.029 (2.257) | 17.736 (2.712)

3. Secondary Outcome: Psychic Anxiety Item of the Hamilton Rating Scale for Depression (HAM-D).
Description: Psychic anxiety item of the Hamilton Rating Scale for Depression (HAM-D) (item 10, 0-4 units), 0 is considered the best outcome.
  Hamilton Rating Scale for Depression (HAM-D)is a 17-item, clinician-rated scale that assesses depressive symptoms. The HAMD-17 consists of 17 symptoms, each of which is rated from 0 to 2 or 0 to 4, where 0 is none/absent. The HAMD-17 total score is calculated as the sum of the 17 individual symptom scores; the total score can range from 0 to 52. Higher HAMD-17 scores indicate more severe depression.
Time Frame: Week 4
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | AZD2327 | Placebo
Number analyzed (Participants) | 13 | 9
Units on a scale | 1.373 (0.313) | 2.128 (0.379)

4. Secondary Outcome: The Number of Participants With at Least 50% Reduction of Hamilton Rating Scale for Depression (HAM-D)Total Score.
Description: Hamilton Rating Scale for Depression (HAM-D) response is defined as a >= 50% reduction from randomization (baseline) in HAM-D total score.
  Hamilton Rating Scale for Depression (HAM-D)is a 17-item, clinician-rated scale that assesses depressive symptoms. The HAMD-17 consists of 17 symptoms, each of which is rated from 0 to 2 or 0 to 4, where 0 is none/absent. The HAMD-17 total score is calculated as the sum of the 17 individual symptom scores; the total score can range from 0 to 52. Higher HAMD-17 scores indicate more severe depression.
Time Frame: Randomization to week 4
Measure: Number; unit: Participants
Arm/Group | AZD2327 | Placebo
Number analyzed (Participants) | 13 | 9
Participants | 5 | 4

5. Secondary Outcome: The Number of Participants With at Least 50% Reduction of Hamilton Rating Scale for Anxiety (HAM-A)Total Score.
Description: Hamilton Rating Scale for Anxiety (HAM-A) response is defined as a >= 50% reduction from randomization (baseline) in HAM-A total score.
  The Hamilton Rating Scale for Anxiety (HAM-A) is used as a rating measure of anxiety severity. The scale consists of 14 items. Each item is rated on a scale of 0 to 4. The HAM-A total score is the sum of the 14 items and the score ranges from 0 to 56, 0 is considered the best outcome.
Time Frame: Randomization to week 4
Measure: Number; unit: Participants
Arm/Group | AZD2327 | Placebo
Number analyzed (Participants) | 13 | 9
Participants | 7 | 3

ADVERSE EVENTS:
Arm/Group | AZD2327 | Placebo
Serious Adverse Events (participants affected / at risk) | 1/13 | 0/9
Other Adverse Events (participants affected / at risk) | 13/13 | 9/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | AZD2327 (N=13) | Placebo (N=9)
Hypotension (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | AZD2327 (N=13) | Placebo (N=9)
Hypotension (Vascular disorders) | 1 | 2
Tachycardia (Cardiac disorders) | 2 | 1
Chest Pain (General disorders) | 6 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Hypertension (Vascular disorders) | 2 | 0
Breast pain (Reproductive system and breast disorders) | 1 | 0
Ear Pain (Ear and labyrinth disorders) | 2 | 1
Tinnitus (Ear and labyrinth disorders) | 5 | 2
Vision blurred (Eye disorders) | 1 | 1
Eye Irritation (Eye disorders) | 2 | 5
Decreased Appetite (Metabolism and nutrition disorders) | 5 | 4
Increased Appetite (Metabolism and nutrition disorders) | 5 | 2
Constipation (Gastrointestinal disorders) | 6 | 4
Diarrhea (Gastrointestinal disorders) | 3 | 2
Flatulence (Gastrointestinal disorders) | 5 | 2
Thirst (General disorders) | 6 | 1
Pollakiuria (Renal and urinary disorders) | 4 | 0
Nausea (Gastrointestinal disorders) | 5 | 2
Abdominal Discomfort (Gastrointestinal disorders) | 6 | 2
Faeces discoloured (Gastrointestinal disorders) | 1 | 0
Dysgeusia (Nervous system disorders) | 4 | 1
Vomiting (Gastrointestinal disorders) | 1 | 1
Weight Increased (Investigations) | 8 | 2
Weight Decreased (Investigations) | 7 | 4
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 | 0
Libido Decreased (Psychiatric disorders) | 3 | 0
Genital Discomfort (Reproductive system and breast disorders) | 1 | 1
Libido Increased (Psychiatric disorders) | 1 | 0
Menstruation Irregular (Reproductive system and breast disorders) | 0 | 1
Dysuria (Renal and urinary disorders) | 0 | 1
Premenstrual syndrome (Reproductive system and breast disorders) | 2 | 0
Dizziness (Nervous system disorders) | 7 | 3
Headache (Nervous system disorders) | 9 | 6
Dental Care (Surgical and medical procedures) | 0 | 2
Dry Mouth (Gastrointestinal disorders) | 9 | 4
Gingival Disorder (Gastrointestinal disorders) | 1 | 1
Salivary Hypersecretion (Gastrointestinal disorders) | 1 | 1
Mouth Ulceration (Gastrointestinal disorders) | 2 | 2
Akathisia (Nervous system disorders) | 0 | 1
Dyskinesia (Nervous system disorders) | 1 | 0
Oedema (General disorders) | 1 | 1
Muscle Rigidity (Musculoskeletal and connective tissue disorders) | 3 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 5 | 3
Tic (Psychiatric disorders) | 1 | 0
Tremor (Nervous system disorders) | 3 | 0
Malignant Dysphagia (Gastrointestinal disorders) | 3 | 0
Influenza (Infections and infestations) | 4 | 1
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 5 | 4
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 4 | 2
Disturbance in attaention (Nervous system disorders) | 2 | 1
Confusional State (Psychiatric disorders) | 1 | 0
Depression (Psychiatric disorders) | 2 | 1
Initial Insomnia (Psychiatric disorders) | 7 | 1
Somnolence (Psychiatric disorders) | 7 | 3
Terminal Insomnia (Psychiatric disorders) | 6 | 2
Hallucinations (Psychiatric disorders) | 1 | 0
Poor quality sleep (Nervous system disorders) | 5 | 3
Irritability (General disorders) | 6 | 3
Memory Impairment (Nervous system disorders) | 3 | 2
Hypokinesia (Psychiatric disorders) | 3 | 0
Psychomotor Hyperactivity (Psychiatric disorders) | 5 | 2
Dysarthria (Nervous system disorders) | 1 | 0
Suicidal Behavior (Psychiatric disorders) | 1 | 0
Suicidal Ideation (Psychiatric disorders) | 2 | 1
Fatigue (General disorders) | 4 | 2
Skin irritation (Skin and subcutaneous tissue disorders) | 4 | 3
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 1
Injury (Injury, poisoning and procedural complications) | 1 | 1
Pyrexia (General disorders) | 2 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No